CLINICAL TRIAL: NCT06882421
Title: Evaluation of the Acceptability and Usability of a Point-of-care-in-vitro Diagnostic Micro-sampling Device for Micronutrient Measurement.
Brief Title: VITAmin and Micronutrient Testing: Acceptability and SCOPE of Point-of-care Device
Acronym: VITASCOPE
Status: Completed | Type: Observational
Sponsor: Norfolk and Norwich University Hospitals NHS Foundation Trust (Other)
Collaborators: University of East Anglia (Other)
Responsible Party: Sponsor
Other Study IDs: Version 1.2 03/06/20; 62431 (Registry Identifier: NIHR Portfolio Study ID)
Record Dates: First submitted 2025-02-25; First posted 2025-03-18 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2024-08

CONDITIONS: Micronutrient Levels
Keywords: micronutrient testing acceptability; Point-of-care device

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Childhood obesity is a global health crisis with 1.2 million children in England severely obese, predisposing them to multiple health risks which decrease lifespan and compromise health. Children suffering from obesity experience a state of paradoxical malnutrition; despite excessive calorie intake they have high rates of micronutrient deficiencies rates due to consumption of energy dense, nutrient poor diets. Around 70-80% of obese children are Vitamin D deficient, 10% have low B12 concentrations and 50% have folic acid deficiency. Currently screening for micronutrient deficiencies does not form a routine part of clinical care at all medical centres because they require a large volume of blood and are expensive to perform. A prototype point-of-care in-vitro diagnostic test has been developed which allows at-home/primary care testing of micronutrient levels, using an integrated finger-prick and minimal amount of blood. This device should be simple to use, with just one push of a button. The results are analysed using a phone app for clear decision-making, with data uploaded to healthcare providers automatically. This study aims to ask service users (young people and their families) for their views on the usability and acceptability of the device prior to developing the product further.

DETAILED DESCRIPTION:
Malnutrition, where there is an insufficient supply or inability to absorb nutrients is classified by the World Health Organisation as the biggest worldwide threat to public health. Untreated malnutrition is an independent risk factor for mortality and is associated with increased healthcare costs. Malnutrition is not only found in association with low weight but is also found in individuals with morbid obesity. Obese individuals experience a state of paradoxical malnutrition; despite excessive dietary intake they have high micronutrient deficiencies rates due to intake of energy-dense, nutrient-poor diets. Childhood obesity is a global health crisis with 1.2 million children in England severely obese, putting them at multiple health risks which lower lifespan and affect health.

Currently micronutrient measurement is performed in hospitals. A large volume (>6mls) is taken with results for some tests taking a minimum of 2 weeks. This delays treatment starting and requires provision of additional clinical time for the results to be fed back to patients and their families. There are significant financial, emotional and carbon costs for patients attending for hospital based blood tests.

A point-of-care blood test for micronutrients has been developed, which uses an integrated finger-prick and minimal amount of blood (40μls). The device is simple to use, with just one push of a button, allowing primary care clinicians and potentially parents/guardians to administer the test.

This study aims to ask young people and their parents/carers for their views on this device before further development is undertaken on the product to ensure it meets with their needs.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged>10 years or parents of a patient being seen in a NNUH CEW clinic.
* Parents/Participants must have capacity to consent/assent and provide a signed and dated informed consent
* Able to participate in an interview regarding the acceptability/usability of the device.

Exclusion criteria:

- Potential participants will not be eligible if they lack capacity to provide informed consent (or in the case of young people under the age of 16, informed assent and informed parental consent)

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 30 children and their parents/carers, attending the Complications of Excess weight (CEW)/ Health Futures Clinic at the Jenny Lind Children's Hospital, NNUH. Parents can participate in the study independently of their children.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2024-06-25 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-09-27 (Actual)

PRIMARY OUTCOMES:
Number of participants and their parents who prefer using a finger prick test for micronutrient measurement. | 12 months
  1. What are the preferences of young people and their families regarding the new technology?
  2. To identify the problems and any benefits of the new technology from patients/parents/guardians/ medical staff

SECONDARY OUTCOMES:
Demographics of study participants | 12 months
  1) Age, gender and ethnicity of participants

CONTACTS AND LOCATIONS:
Overall Officials: Emma Webb, PhD, Principal Investigator — Consultant at NNUH
Locations (1):
- Norfolk and Norwich University Hospitals NHS Foundation Trust, Norwich, Norfolk, United Kingdom

IPD SHARING:
Plan to Share IPD: No